CLINICAL TRIAL: NCT03224585
Title: Treatment of Acute Pericarditis With Anakinra
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was terminated because dramatic benefits seen during the first 24 hours of drug administration combined with COVID restrictions on research activities suggested it was both unethical and unnecessary to complete the planned enrollment
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HM20008638
Record Dates: First submitted 2017-07-19; First posted 2017-07-21 (Actual); Results first posted 2021-02-23 (Actual); Last update posted 2021-02-23 (Actual); Status verified 2021-02

CONDITIONS: Acute Pericarditis
Keywords: anakinra; Kineret; pericarditis
MeSH Terms: conditions — Pericarditis | interventions — Interleukin 1 Receptor Antagonist Protein

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Anakinra (Experimental): 100 mg subcutaneous injection
  Interventions: Drug: Anakinra
- Placebo (Placebo Comparator): 100 mg NaCl 0.9% subcutaneous injection
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Anakinra — Period 1 (Time 0-72 hours) - this will be an open-label phase during which all subjects meeting enrollment criteria will receive anakinra 100 mg subcutaneously injections daily for 3 days.
  Period 2 (Time 72 hours to 7 days) - anakinra 100 mg subcutaneous injections daily for 4 days
  Arms: Anakinra
Drug: Placebo — Period 1 (Time 0-72 hours) - this will be an open-label phase during which all subjects meeting enrollment criteria will receive anakinra 100 mg subcutaneously injections daily for 3 days.
  Period 2 (Time 72 hours to 7 days) - placebo 100 mg saline subcutaneous injections daily for 4 days
  Arms: Placebo

SUMMARY:
The goal of this study is to determine the safety and efficacy of anakinra for the treatment of acute pericarditis when initiated within 6 hours of diagnosis and continued for 3 or 7 days.

1. to determine the efficacy of anakinra with respect to chest pain resolution
2. to determine the safety of anakinra with respect to adverse drug events

DETAILED DESCRIPTION:
Acute pericarditis is a clinical syndrome characterized by a profound inflammation of the membrane tissue that surrounds, supports and protects the heart. Acute pericarditis can be caused by a variety of infectious and non-infectious agents, but it most commonly either follows a viral infection of the upper respiratory tract or has no apparent cause.

Acute pericarditis occurs rather abruptly in previously healthy individuals, generally a child or young adult. Most cases of acute pericarditis resolve within a few days with non-steroidal anti-inflammatory drugs. However, patients experience severe chest pain and are at high risk for life-threatening complications involving the pericardium, such as pericardial tamponade. Acute pericarditis is diagnosed in 1 in 20 (5%) ED visits for chest pain.

Anakinra (Kineret) has been shown to treat and cure refractory and recurrent pericarditis. This study is aimed at determining whether anakinra is also effective as first line treatment in acute pericarditis.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥12 years in presence of a parent able to provide consent or age >18 years
* First or recurrent episode of acute pericarditis, defined as the presence of at least 2 of the following:
* Chest pain (suggestive of pericarditis and not explained by another condition)
* Pericardial friction rub on physical exam
* ST-segment elevation and/or PR depression on ECG
* New or worsening pericardial effusion
* Pain of moderate-to-severe intensity (pain score ≥6 on a scale of 0-10 where 0 is no pain at all and 10 is the worst pain ever experienced) at time on enrollment
* Ability to provide written informed consent if 18 years or older or to provide assent in presence of parental consent if 12-17 years of age

Exclusion Criteria:

* Pericarditis due to known bacterial or fungal infection
* Pericarditis due to known malignancy
* Pericarditis after cardiac surgery
* Tamponade or need for pericardiocentesis for diagnostic/therapeutic purposes
* Pregnancy or breastfeeding
* Hypersensitivity to anakinra, latex or products derived from Escherichia coli
* Chronic pain syndrome or chronic use of analgesic drugs

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2018-05-11 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2020-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Abbate, MD, PhD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

REFERENCES:
- [Derived] Wohlford GF, Buckley LF, Vecchie A, Kadariya D, Markley R, Trankle CR, Chiabrando JG, de Chazal HM, Van Tassell B, Abbate A. Acute Effects of Interleukin-1 Blockade Using Anakinra in Patients With Acute Pericarditis. J Cardiovasc Pharmacol. 2020 Jul;76(1):50-52. doi: 10.1097/FJC.0000000000000847. PMID 32398478

RESULTS

PARTICIPANT FLOW:
Groups:
- Anakinra (3 Days) Then Anakinra (4 Days): Period 1 (Time 0-72 hours) - this will be an open-label phase during which all subjects meeting enrollment criteria will receive anakinra 100 mg subcutaneously injections daily for 3 days.
  Period 2 (Time 72 hours to 7 days) - anakinra 100 mg subcutaneous injections daily for 4 days
- Anakinra (3 Days) Then Placebo (4 Days): Period 1 (Time 0-72 hours) - this will be an open-label phase during which all subjects meeting enrollment criteria will receive anakinra 100 mg subcutaneously injections daily for 3 days.
  Period 2 (Time 72 hours to 7 days) - placebo 100 mg saline subcutaneous injections daily for 4 days
Period: Overall Study
Arm/Group | Anakinra (3 Days) Then Anakinra (4 Days) | Anakinra (3 Days) Then Placebo (4 Days)
Started | 2 | 3
Completed | 2 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Anakinra (3 Days) Then Anakinra (4 Days): 100 mg subcutaneous injection
  Anakinra: Period 1 (Time 0-72 hours) - this will be an open-label phase during which all subjects meeting enrollment criteria will receive anakinra 100 mg subcutaneously injections daily for 3 days.
  Period 2 (Time 72 hours to 7 days) - anakinra 100 mg subcutaneous injections daily for 4 days
- Anakinra (3 Days) Then Placebo (4 Days): 100 mg NaCl 0.9% subcutaneous injection
  Placebo: Period 1 (Time 0-72 hours) - this will be an open-label phase during which all subjects meeting enrollment criteria will receive anakinra 100 mg subcutaneously injections daily for 3 days.
  Period 2 (Time 72 hours to 7 days) - placebo 100 mg saline subcutaneous injections daily for 4 days
- Total: Total of all reporting groups
Arm/Group | Anakinra (3 Days) Then Anakinra (4 Days) | Anakinra (3 Days) Then Placebo (4 Days) | Total
Number analyzed (Participants) | 2 | 3 | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 3 | 5
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 42 (9) | 40 (16) | 41 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 1 | 3 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 1 | 2 | 3
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 2 | 3 | 5

OUTCOME MEASURES:

1. Primary Outcome: Pain Score
Description: Change from baseline in visual analog pain score from 0 to 10.
  For this visual analog pain scale, the patient is asked to rate their pain from 0 to 10. A score of 0 represents "no pain", a score of 5 represents "moderate pain", and 10 represents "worst pain".
Time Frame: Baseline to 6 hours
Measure: Median (Inter-Quartile Range); unit: units on a scale
Groups:
- All Patients: This group includes all patients enrolled in the clinical trial
Arm/Group | All Patients
Number analyzed (Participants) | 5
units on a scale | -3 [-3 to -2]
Statistical Analysis 1: Comparison: All Patients; This analysis compared the change in pain scores between baseline and 6 hours; Test type: Superiority; p = 0.0121, Paired samples Wilcoxon test

2. Secondary Outcome: Pain Score
Description: as for outcome 1
Time Frame: Baseline to 24 hours
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | All Patients
Number analyzed (Participants) | 5
units on a scale | -4 [-4.25 to 4]
Statistical Analysis 1: Comparison: All Patients; Test type: Superiority; p = 0.0025, Paired samples Wilcoxon test

ADVERSE EVENTS:
Time Frame: 30 days
Description: Adverse events assessed via daily physician examination and routine labs
Arm/Group | Anakinra (3 Days) Then Anakinra (4 Days) | Anakinra (3 Days) Then Placebo (4 Days)
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/2 | 3/3
Other Adverse Events (participants affected / at risk) | 1/2 | 1/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Anakinra (3 Days) Then Anakinra (4 Days) (N=2) | Anakinra (3 Days) Then Placebo (4 Days) (N=3)
Thrombophlebitis - After completion of anakinra (Vascular disorders) | 0 (0) | 1 (1)
Coronary vasospasm - After completion of anakinra (Cardiac disorders) | 0 (0) | 1 (1)
Resistant pericarditis - After completion of anakinra (Cardiac disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Anakinra (3 Days) Then Anakinra (4 Days) (N=2) | Anakinra (3 Days) Then Placebo (4 Days) (N=3)
Injection site reactions - While taking anakinra (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Informed Consent Form (2017-06-08): https://cdn.clinicaltrials.gov/large-docs/85/NCT03224585/ICF_000.pdf
  • Study Protocol (2017-06-08): https://cdn.clinicaltrials.gov/large-docs/85/NCT03224585/Prot_001.pdf
  • Statistical Analysis Plan (2017-06-08): https://cdn.clinicaltrials.gov/large-docs/85/NCT03224585/SAP_002.pdf